CLINICAL TRIAL: NCT01851382
Title: Collection of Saliva and/ or Peripheral Blood From Healthy Volunteers for Research
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130128; 13-C-0128
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Graft vs Host Disease; Healthy Volunteer; Graft-Versus-Host Disease
Keywords: ELISA; Spectrometry; Protein Biomarkers; Proteomic Analyses; Natural History
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Healthy volunteers.

SUMMARY:
Background:

- Researchers often collect samples from healthy volunteers to further their research. These samples can help better understand serious side effects and complications of transplant treatments in patients. This study will collect saliva samples from healthy volunteers.

Objectives:

- To collect saliva and blood samples from healthy volunteers for research studies.

Eligibility:

- Healthy men ages 30-70 years for Phase I of the study.

Design:

* Participants will be screened with a medical history questionnaire. They will also have a brief oral exam to check for any mouth infection.
* Participants will provide a saliva sample. The collection process will take about 5 minutes.
* No treatment will be given as part of this study.

DETAILED DESCRIPTION:
Background:

* Chronic graft-versus-host disease (cGVHD) is a severe immunological complication that occurs after allogeneic hematopoietic stem cell transplantation (HSCT). Although oral cGVHD occurs in >25% of cGVHD patients and leads to decreased quality of life, its etiology is poorly understood.
* The primary objective of the present protocol is to enroll normal volunteers who will contribute a saliva and/or blood sample in order to compare its characteristics with those of patients with and without chronic GVHD after allogeneic HSCT. The normal control saliva and blood samples will provide a standard of comparison for patient saliva and blood samples from ongoing NCI cGVHD related protocols.

Objective:

-To collect approximately 5 ml of saliva and/or 18 cc peripheral blood from healthy volunteers as needed to support research activities.

Eligibility:

* Healthy individuals (including employees) all racial/ethnic groups, aged 18 years or older.
* Volunteers must be willing to undergo saliva and peripheral blood collection.
* No active illnesses, immunodeficiency, history of opportunistic infection, autoimmune disease, immunosuppressive medications or prior organ, bone marrow or peripheral blood stem cell transplant.
* Ability of subject to understand and provide written informed consent.
* Phase I of the study will be restricted to males, age 30-70 years

Design:

* Healthy volunteers will be offered the opportunity to participate in this protocol.
* A basic clinical dental assessment will be done.
* Saliva samples will be collected from the consenting subject.
* Peripheral blood samples may be collected from the consenting subject at the same visit.
* Protein assays will be performed on the collected saliva and blood samples.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy individuals (including employees) and other healthy volunteers from all racial/ethnic groups
* Age 18 years and older, with possible restriction for age-matching to patient samples.
* Ability of subject to understand and provide written informed consent
* Subjects must participate fully and be willing to comply with the procedures of the protocol
* Phase I of the study will be restricted to males, age 30-70 years.

EXCLUSION CRITERIA:

* Active systemic illnesses, immunodeficiency, history of opportunistic infection, autoimmune disease, immunosuppressive medications
* Prior organ, bone marrow or peripheral blood stem cell transplant
* Acute dental infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers from the local community.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2015-02-12 (Actual)

PRIMARY OUTCOMES:
Collect saliva and peripheral blood | End of specimen collection
  Sample analysis for research.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mays JW, Fassil H, Edwards DA, Pavletic SZ, Bassim CW. Oral chronic graft-versus-host disease: current pathogenesis, therapy, and research. Oral Dis. 2013 May;19(4):327-46. doi: 10.1111/odi.12028. Epub 2012 Oct 28. PMID 23107104
- [Background] Bassim CW, Ambatipudi KS, Mays JW, Edwards DA, Swatkoski S, Fassil H, Baird K, Gucek M, Melvin JE, Pavletic SZ. Quantitative salivary proteomic differences in oral chronic graft-versus-host disease. J Clin Immunol. 2012 Dec;32(6):1390-9. doi: 10.1007/s10875-012-9738-4. Epub 2012 Jul 18. PMID 22806177
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0128.html